CLINICAL TRIAL: NCT07021001
Title: Prevention and Promotion of Mental Well-being in Adolescents: Efficacy of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders as a School-based Universal Prevention Program (UP-A Kind) Through a Cluster Randomized Controlled-trial
Brief Title: Promotion of Mental Health in Adolescents: A School-Based Preventive Version of the Unified Protocol (UP-A Kind)
Acronym: UP-A Kind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: EPIS Association - Entrepreneurs for Social Inclusion (Unknown); Z Zurich Foundation (Unknown); Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Inês Maçãs de Carvalho, MSc, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022.154441.BD
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: The Focus is the Prevention and Promotion of Mental Well-being and is a Universal Delivery Intervention
Keywords: Mental Well-being; Unified Protocol; Adolescents; Transdiagnostic Processes; Emotion Regulation; Universal prevention; School
MeSH Terms: conditions — Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This is longitudinal research. The Cluster Randomized Control Trial include a Control Group (N=150) and an Experimental Group (N=150).
Who Masked: Participant
Masking Description: Baseline assessment occurs previously to allocation to experimental and control groups. Outcomes assessor is blind to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): UP-A Kind is a school based universal preventive intervention with 8 sessions adapted from the UP-A. Intervention is delivered in eight weekly sessions (each session lasting around 100 minutes). Participants pertaining to this group will be assessed at 4 different time points (pre- and post-treatment and at a 3-, 6- and 12- month follow-up).
  Interventions: Behavioral: UP-A, a cognitive-behavioral structured group intervention, was adapted as a universal preventive intervention to be delivered in school settings (UP-A Kind).
- Control Group (No Intervention): Control group participants will receive no treatment and will be assessed at the same time points as participants from the Experimental group (pre- and pos-intervention, 3-, 6- and 12-month follow-up). Participants in Control group will be offered the possibility of participating in the UP-A Kind after the 12-month follow-up in a voluntary basis. Nevertheless, data from this delivery will not be included in the clinical trial.

INTERVENTIONS:
Behavioral: UP-A, a cognitive-behavioral structured group intervention, was adapted as a universal preventive intervention to be delivered in school settings (UP-A Kind). — The UP-A Kind is a school-based universal prevention intervention that aims to promote adaptive emotion regulations strategies, enhance mental well-being and prevent emotional disorders with the following contents: motivating to take care of mental well-being, psychoeducation about emotions, awareness of physical sensations, cognitive lexibility, behavioral experiences, recognizing warning signs, and promoting a compassionate attitude towards the self and others.
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to assess the efficacy of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders for Adolescents (UP-A; Ehrenreich-May et al., 2018) as a universal school-based preventive intervention (UP-A Kind) in adolescents aged 11-18. This intervention aims to prevent emotional symptoms and improve adolescents' mental well-being in school setting, assessing changes in transdiagnostic processes. Researchers will compare an experimental group and a control group. Participants will participate in eight weekly sessions and will be assessed at 4 time points (pre- and post-treatment and 3-, 6- and 12-month follow-up). Control group participants will receive no intervention and will be assessed at the same time points.

DETAILED DESCRIPTION:
Emotional disorders are highly prevalent during adolescence, and significantly impact the development and well-being of adolescents. The World Health Organization defines preventive interventions and promotion of adolescent mental health as a priority. Nevertheless, many adolescents lack access to psychological interventions, leading to short, medium, and long-term impacts. The school setting is a privileged context for the implementation of universal preventive interventions as it offers accessibility to all adolescents. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A; Ehrenreich-May et al., 2018), a transdiagnostic intervention, has demonstrated effectiveness in reducing anxiety and depressive symptoms and improving quality of life in this population. Preventive transdiagnostic interventions may have better results in the long term. The main goal is to assess the efficacy of UP-A as a preventive intervention. The goal is prevent emotional symptoms and improve mental well-being, assessing changes in transdiagnostic factors, including cognitive flexibility, mindfulness, and distress tolerance. Participants are adolescents aged 11-18 that frequent 7-9 grade. The intervention will be delivered by clinical psychologists. The design is a cluster randomized controlled trial with two groups: control group and experimental group. Pre- and post-intervention, and follow-up at 3, 6 and 12 months will be carried out.

All procedures were approved by the Ethics Committee of the Faculty of Psychology and Educational Sciences, University of Coimbra and the School Boards authorized the data collection protocol to be implemented in school contexts. Informed consent from adolescents and their parents/legal guardians will be required. Adolescents and their parents/legal guardians will be informed that the participation is voluntary, confidential and that they can decline to participate at any time without any consequence.

ELIGIBILITY:
Inclusion Criteria:

* Frequent 7º, 8º or 9º grade
* Providing written informed assent (the adolescent and the legal tutor)
* Being able to understand, write and read Portuguese

Exclusion Criteria:

* No exclusion criteria because of being a universal prevention study

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Socio-Demographic Information Questionnaire | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
Mental Health Continuum-Short Form (Keyes et al., 2008) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure Positive Mental Health.
Kidscreen-10 (Portuguese version: Matos et al., 2012) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure quality of life.
Overall Depression Severity and Impairment Scale (ODSIS) (Bentley, Gallagher, Carl, Barlow, 2014) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  ODSIS was used to measure Depression and was translate and adapt to Portuguese for this study.
Overall Anxiety Severity and Impairment Scale (OASIS) (Norman, Cissell, Means-Christensen, & Stein, 2006) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  OASIS was used to measure Anxiety and was translate and adapt to Portuguese for this study.
School Connectedness Scale (SCS) (Furlong and O'Brennan, 2011) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure School connectedness and was adapted and translated to Portuguese for this study.

SECONDARY OUTCOMES:
Social Emotional Abilities Survey (UNICEF, 2023) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was adapted and translated to Portuguese for this study.
The Multidimensional Emotional Disorder Inventory (MEDI) (Rosellini & Brown, 2019) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure transdiagnostic dimensions of Emotional disorders.
Difficulties in Emotion Regulation Scale Short Form (DERS-SF) (Portuguese version: Moreira et al., 2020) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure emotion regulation difficulties.
Emotional Avoidance Strategy Inventory for Adolescents (EASI-A) (Kennedy & Ehrenreich-May, 2016) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  This measure is an adaptation of an adult measure of emotional avoidance (Fairholme, Ehrenreich-May, Ellard, Boisseau, Farchione, Barlow, 2008) and was adapted and translated to Portuguese for this study.
Distress Tolerance Scale (DTS) (Tonarely & Ehrenreich-May, 2020) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure distress tolerance.
Child and Adolescent Mindfulness Measure (CAMM) (Portuguese version: Cunha et al., 2013) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure Mindfulness.
Self-Compassion Scale (SCS) (Portuguese version: Cunha et al., 2016) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure self-compassion.
Social Safeness and Pleasure Scale (SSPS-A) (Gilbert et al., 2009) | Baseline, Week 8, Follow-Up 3 Months, Follow-Up 6 Months and Follow-Up 12 Months
  The scale was used to measure Social Safeness.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC), Faculty of Psychology and Educational Sciences - University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided